CLINICAL TRIAL: NCT05012501
Title: Analysis of Neutrophil Extracellular Traps in Hypercoagulability and Portal Vein Thrombosis in Liver Cirrhosis Patients
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYWZLL26363
Record Dates: First submitted 2021-07-15; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Neutrophil Extracellular Trap Formation; Portal Vein Thrombosis; Liver Cirrhosis
Keywords: Neutrophil Extracellular Trap Formation; Portal Vein Thrombosis; Hypercoagulability
MeSH Terms: conditions — Liver Cirrhosis; Thrombophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: None Retained — Plasm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PVT group: （1) Patients with cirrhosis diagnosed in accordance with the 2019 Guidelines for the Diagnosis and Treatment of Cirrhosis;(2) In accordance with the diagnostic criteria of portal vein thrombosis in the 2015 European Society of Hepatology Clinical Practice Guidelines: Hepatic Vascular Diseases. Color ultrasound, CT, MRI, and other imaging studies confirmed the presence of portal vein thrombosis and the specific location of the thrombosis.
  Interventions: Diagnostic Test: test NETs markers
- without PVT group: (1) Patients with cirrhosis diagnosed in accordance with the 2019 Guidelines for the Diagnosis and Treatment of Cirrhosis;(2)Color ultrasound, CT, MRI, and other imaging studies confirmed the absence of portal vein thrombosis and the specific location of the thrombosis.
  Interventions: Diagnostic Test: test NETs markers

INTERVENTIONS:
Diagnostic Test: test NETs markers — NETs markers (Myeloperoxidase, Neutrophil elastase, Citrate histone H3), tissue factor, endotoxin, factor X, TAT complex, and anti-β2 glycoprotein I were detected in plasma using capture ELISA and specific ELISA kits.

SUMMARY:
The aim of this study was to investigate whether NETs markers can enhance procoagulant activity and predict portal vein thrombosis in patients with live cirrhosis, so as to establish a novel predictor to guide clinical decision-making.So we recruit liver cirrhosis with portal vein thrombosis and without portal vein thrombosis treated at the Affiliated Hospital of Qingdao University and collection of blood samples.

DETAILED DESCRIPTION:
Seventy-nine patients with benign liver cirrhosis treated at the Affiliated Hospital of Qingdao University (China) from September 2020 to January 2021 were recruited for this study, including 26 patients with portal vein thrombosis and 53 patients without portal vein thrombosis. NETs markers (Myeloperoxidase, Neutrophil elastase, Citrate histone H3), tissue factor, endotoxin, factor X, TAT complex, and anti-β2 glycoprotein I were detected in plasma using capture ELISA and specific ELISA kits. T-test was performed to analyze whether there was a statistical difference between the two groups, and regression analysis was performed between NETs markers and tissue factor, endotoxin, factor X, TAT complex, and anti-β2 glycoprotein I to investigate whether there was a correlation. This study without any intervention measures, will not cause harm.

ELIGIBILITY:
Inclusion Criteria:

（1) Clinical diagnosis of liver cirrhosis (2) Clinical diagnosis of portal vein thrombosis

Exclusion Criteria:

1. primary or secondary liver malignancy
2. hematologic diseases
3. Bud-Chiah syndrome
4. incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Seventy-nine patients with benign liver cirrhosis treated at the Affiliated Hospital of Qingdao University (China) from September 2020 to January 2021 were recruited for this study, including 26 patients with portal vein thrombosis and 53 patients without portal vein thrombosis.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Concentration of NETs markers | 1 year.
  NETs markers (Myeloperoxidase, Neutrophil elastase, Citrate histone H3), tissue factor, endotoxin, factor X, TAT complex, and anti-β2 glycoprotein I were detected in plasma using capture ELISA and specific ELISA kits.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided